CLINICAL TRIAL: NCT03793192
Title: Promoting Activity After COPD Exacerbations, Aim 2 (PACE2)
Brief Title: Promoting Activity After COPD Exacerbations, Aim 2
Acronym: PACE2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution, data collected is insufficient for analysis
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jerry Krishnan, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-1526; 5K23HL130524-03 (NIH)
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Intervention versus Enhanced Usual Care
Who Masked: Outcomes Assessor
Masking Description: Allocation sequence will be concealed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PACE2 Intervention (Experimental): All participants will receive usual healthcare as per their treating medical team and carry a pedometer for recording of physical activity. In addition, participants randomized to the PACE2 intervention will receive written educational materials regarding physical activity, telephone-based coaching to integrate physical activity in daily life activities and address barriers to attending pulmonary rehabilitation.
  Interventions: Other: PACE2 Intervention
- Enhanced Usual Care (No Intervention): All participants will receive usual healthcare as per their treating medical team and carry a pedometer for recording of physical activity.

INTERVENTIONS:
Other: PACE2 Intervention — Written educational materials regarding physical activity, telephone-based coaching to integrate physical activity in daily life activities and address barriers to attending pulmonary rehabilitation.
  Arms: PACE2 Intervention

SUMMARY:
This randomized controlled pilot study involving patients with chronic obstructive pulmonary disease (COPD) recently discharged from the hospital will evaluate the feasibility and efficacy of a home-based mobile-health supported physical activity promotion program.

DETAILED DESCRIPTION:
Deconditioning is common in patients with chronic obstructive pulmonary disease (COPD) and has been associated with poor outcomes (e.g. difficulty breathing). Pulmonary rehabilitation (PR) initiated shortly after hospital discharge following a COPD exacerbation has been shown to improve some of these outcomes. However, for many patients, access to PR programs is limited due to environmental, physical, and psycho-social reasons. Home-based physical activity promotion, combined with education and social support, could help to overcome some barriers to access and have been shown to be effective in populations with mild to moderate COPD. However, home-based interventions have not been tested in patients recovering from COPD exacerbations, a group for whom solutions to safely promote physical activity are urgently needed. In PACE2 up to 64 adult participants with a physician diagnosis of COPD will be enrolled and randomized to one of two groups: physical activity promotion intervention or enhanced usual care. Participants will be enrolled while hospitalized and randomization will occur approximately 7 days after hospital discharge. All participants will be provided self-management educational materials and community resources both prior to hospital discharge and during a home visit shortly after hospital discharge. For the participants randomized to the intervention group, physical activity promotion will start following randomization and continue for 12 weeks. These participants will also receive a personalized plan to attend pulmonary rehabilitation, a guideline-recommended program for patients with COPD recovering from exacerbations. The primary endpoint will be the change in physical activity (mean daily step counts over 1 week) over time using repeated measures over the 12 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Physician diagnosis of COPD;
3. Hospitalized as an inpatient, 23-hour observation, or clinical decision unit
4. Admitting respiratory conditions sensitive to the Centers for Medicare and Medicaid Services Hospital Readmission Reduction Program as listed below:

   * COPD exacerbation
   * Asthma/COPD overlap
   * Decompensated heart failure
   * Pneumonia
   * Chronic Airway Disease

Exclusion Criteria:

1. Physical inability to participate in a walking program;
2. Oxygen saturation <90% by pulse oximetry refractory to supplemental oxygen, or in a patient unable or unwilling to use supplemental oxygen;
3. Fall in the previous 6 months;
4. Resting electrocardiogram (ECG) with new ST changes or tachyarrhythmia;
5. Planned discharge home to hospice or to long term care facility/skilled nursing facility;
6. Life expectancy <3 months;
7. Medical contraindication to participating in a physical activity promotion program as determined by the inpatient treating clinician;
8. Unable to communicate in English;
9. Unable or declines to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Change in mean daily step counts | 12 weeks
  change in mean daily step counts (averaged over 1 week) over time using repeated measures over the 12 weeks of the study.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Depression | 12 weeks
  Change in T-score from baseline to week 12 (A negative change in score indicates less emotional distress - depression).
PROMIS Emotional Distress - Anxiety | 12 weeks
  Change in T-score from baseline to week 12 (A negative change in score indicates less emotional distress - anxiety).
PROMIS Fatigue | 12 weeks
  Change in T-score from baseline to week 12 (A negative change in score indicates less fatigue).
PROMIS Physical function | 12 weeks
  Change in T-score from baseline to week 12 (A negative change in score indicates lower physical function).

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Krishnan, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No